CLINICAL TRIAL: NCT02544542
Title: A Comparative Clinical Trial of a New Rectum Cooling System Versus Temperature-adjusting Blanket on Patients of Hypoxic-ischemic Brain Damage
Brief Title: Clinical Trial of a New Rectum Cooling System on Patients of Hypoxic-ischemic Brain Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Collaborators: Chongqing Science and Technology Commission (Other)
Responsible Party: Principal Investigator, Zelan Zuo, Head Nurse of Pediatric Intensive Care Unit, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: X3348
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Mild Hypothermia; Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rectum cooling system (Experimental): Insert the self-made device into the patient's rectum, pump ice-cold saline in to induce mild hypothermia, sustain the desired temperature for 12 hours,then let the body rewarm slowly. Body temperature changes are achieved by controlling the pumping speed of saline.
  Interventions: Device: Rectum cooling system
- Hyper-hypothermia blanket (Active Comparator): Let the patient sleep on the hyper-hypothermia blanket, set the target temperature to induce mild hypothermia, sustain the desired temperature for 12 hours,then let the body rewarm slowly. Body temperature changes are achieved by adjusting the target temperature of the device accordingly.
  Interventions: Device: Hyper-hypothermia blanket

INTERVENTIONS:
Device: Rectum cooling system
  Arms: Rectum cooling system
Device: Hyper-hypothermia blanket
  Arms: Hyper-hypothermia blanket

SUMMARY:
This study will try to evaluate the effectiveness and safety of a new method for achieving mild hypothermia, i.e.,mild hypothermia therapy through rectum. Half of participants will be treated by the widely-used hyper-hypothermia blanket method, while the other half will be treated by the investigators' new method.

DETAILED DESCRIPTION:
Mild hypothermia therapy has been proved to be beneficial to patients with severe traumatic brain injury. Currently a variety of cooling methods can achieve mild hypothermia,the hyper-hypothermia blanket being the most widely-used one.

Hyper-hypothermia blanket is a waterbed mattress connected to a thermostat-controlled water tank. Water is cooled in the tank and recycled between the tank and the mattress so that the patients sleeping on the mattress can be stably cooled. The operation is basically program-controlled ,but the whole system is quite expensive.

The investigators came up with a new cooling system which is very simple and accessible. A condom inserted with two 10# gastric tube and one 6# gastric tube and ringed with a rubber band is inserted into the patient's rectum, and ice-cold saline is pumped in through one 10# gastric tube and drained out from the other 10# gastric tube, the 6# gastric tube connected to the pressure monitor. Cooling rate is controlled by the flow speed of cold saline. The investigators will evaluate the effectiveness and safety of this new method for achieving mild hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal HIE
* After cardiopulmonary resuscitation (CPR)
* Severe craniocerebral injury (GCS < 8)
* Acute central nervous system infection and severe brain edema or lasting convulsion
* Severe cerebral edema caused by various metabolic factors

Exclusion Criteria:

* End-stage heart failure
* Uncorrected serious cardiovascular dysfunction
* Active intracranial hemorrhage not under control
* Platelet count < 50 * 10^9 / L

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Rate of Cooling | 4 hours
  The body temperature is measured every 15 minutes until the target temperature(33-35℃)is reached.
Body Temperature Fluctuations in Maintenance Phase | 12 hours
  During the maintenance phase,the body temperature is measured every 15 minutes.
Rate of Rewarming | 24 to 48 hours
  The body temperature is measured every 15 minutes until it rises to 36.5℃.

SECONDARY OUTCOMES:
Incidence of Complications | 24 to 72 hours
  Any occurence of shiver，arrhythmia and coagulation abnormalities during the therapy.
Fecal Occult Blood Testing Results Before and After the Therapy | Within 24 hours before the therapy and 48 to 72 hours after the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zelan Zuo, Bachelor, Principal Investigator — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Polderman KH, Herold I. Therapeutic hypothermia and controlled normothermia in the intensive care unit: practical considerations, side effects, and cooling methods. Crit Care Med. 2009 Mar;37(3):1101-20. doi: 10.1097/CCM.0b013e3181962ad5. PMID 19237924
- [Background] Polderman KH. Mechanisms of action, physiological effects, and complications of hypothermia. Crit Care Med. 2009 Jul;37(7 Suppl):S186-202. doi: 10.1097/CCM.0b013e3181aa5241. PMID 19535947
- [Background] Badjatia N, Strongilis E, Prescutti M, Fernandez L, Fernandez A, Buitrago M, Schmidt JM, Mayer SA. Metabolic benefits of surface counter warming during therapeutic temperature modulation. Crit Care Med. 2009 Jun;37(6):1893-7. doi: 10.1097/CCM.0b013e31819fffd3. PMID 19384208
- [Background] Thoresen M, Satas S, Loberg EM, Whitelaw A, Acolet D, Lindgren C, Penrice J, Robertson N, Haug E, Steen PA. Twenty-four hours of mild hypothermia in unsedated newborn pigs starting after a severe global hypoxic-ischemic insult is not neuroprotective. Pediatr Res. 2001 Sep;50(3):405-11. doi: 10.1203/00006450-200109000-00017. PMID 11518829
- [Background] Steiner T, Friede T, Aschoff A, Schellinger PD, Schwab S, Hacke W. Effect and feasibility of controlled rewarming after moderate hypothermia in stroke patients with malignant infarction of the middle cerebral artery. Stroke. 2001 Dec 1;32(12):2833-5. doi: 10.1161/hs1201.99511. PMID 11739982